CLINICAL TRIAL: NCT02930824
Title: Implementing Genomics in Practice (IGNITE) Proof of Concept Study: CYP2C19 Genotype-supported Versus Conventional Proton Pump Inhibitor Dosing
Brief Title: Genotype-supported Versus Conventional Proton Pump Inhibitor Dosing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Nemours Children's Hospital (Other); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB201601774-N; U01HG007269 (NIH)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adult Genotype guided treatment (Experimental): For adults randomized to the genotype-supported arm a CYP2C19 genotype will be provided to physicians to assist in dosing.
  Interventions: Genetic: CYP2C19 genotyping
- Adult Conventional treatment (No Intervention): For adults randomized to the conventional arm no genotype will be provided to physicians to assist in dosing.
- Pediatric Genotype guided treatment (Experimental): For children randomized to the genotype-supported arm a CYP2C19 genotype will be provided to physicians to assist in dosing.
  Interventions: Genetic: CYP2C19 genotyping
- Pediatric Conventional treatment (No Intervention): For children randomized to the conventional arm no genotype will be provided to physicians to assist in dosing.

INTERVENTIONS:
Genetic: CYP2C19 genotyping — All proton pump inhibitors are metabolized in part by the CYP2C19 enzyme, which is encoded by the highly polymorphic CYP2C19 gene. Based on variations within this gene the effectiveness of the drug may be reduced.
  Arms: Adult Genotype guided treatment; Pediatric Genotype guided treatment

SUMMARY:
Investigators will conduct a comparative effectiveness study of genotype-supported vs. conventional PPI dosing. Adults and children presenting with Gastroesophageal Reflux Disease (GERD) or dyspepsia symptoms and either 1) being initiated on proton pump inhibitor (PPI) therapy or 2) with continued symptoms on current PPI therapy will be recruited from gastroenterology clinics and randomized to a genotype-supported versus conventional PPI therapy management strategy.

DETAILED DESCRIPTION:
The efficacy of proton pump inhibitors (PPIs) is highly dependent on plasma concentrations achieved following drug administration. All PPIs are metabolized in part by the CYP2C19 enzyme, which is encoded by the highly polymorphic CYP2C19 gene. Depending on the CYP2C19 genotype, individuals are classified into different metabolizer phenotypes: poor metabolizers (PM, 2 loss-of-function CYP2C19 alleles); intermediate metabolizers (IM, one loss-of-function allele); normal metabolizers (NM, no loss or gain-of-function alleles); rapid metabolizer (RM; one gain-of-function allele) and ultra-rapid metabolizers (UM, two gain-of function-alleles). Genetic variants in CYP2C19 are known to profoundly influence PPI plasma concentrations and consequently, response to PPI therapy. For example, individuals classified as either RM or UM have lower PPI concentrations compared to NM or loss-of-function (LOF) allele carriers, respond poorly to PPI therapy, and some fail to respond even when the PPI dose is increased. The investigators hypothesize that genotype-supported PPI dosing will lead to better GERD control and improvement in severity of dyspepsia symptoms compared to conventional dosing. The investigators will conduct a comparative effectiveness study of genotype-supported vs. conventional PPI dosing. Patients presenting with GERD or dyspepsia symptoms and either 1) being initiated on PPI therapy or 2) with continued symptoms on current PPI therapy will be recruited from gastroenterology clinics and randomized to a genotype-supported versus conventional PPI therapy management strategy. The investigators will integrate individual CYP2C19 genotype information into dosing decisions for the genotype-supported arm and compare change in symptom control from baseline to the end of the study between study arms. Given that PPI efficacy is related to PPI exposure and to metabolizer phenotype, individualizing treatment using CYP2C19 genotype-supported dosing is expected to improve symptom management. The investigators will also evaluate patient and clinician knowledge and attitudes about pharmacogenetics testing and physician acceptance of genetic information into clinical practice. Finally, the investigators will collect preliminary data on the potential impact of CYP2C19-supported PPI dosing on adverse event rates.

ELIGIBILITY:
Pediatric:

Inclusion Criteria:

* 5-17 years of age
* diagnosed with GERD or any other stomach acid mediated condition for which a PPI treatment is provided
* currently under a Proton Pump Inhibitor (PPI) therapy or will start a PPI therapy
* Parents/legal guardians and or child must have access to internet and a valid email address

Exclusion Criteria:

* history of extensive esophageal or gastric surgery
* diagnosed with any major chronic illness or conditions that in the opinion of the gastroenterologist that would interfere with participation in the study
* history of Phenylketonuria (PKU) and patients with a history of previous adverse effects from PPI treatment or sensitivity to aspartame (NutraSweet, Equal)

Adult:

Inclusion Criteria:

* 18 years of age or older
* Gastroesophageal Reflux Disease symptoms
* Being initiated on PPI therapy OR continues to have symptoms despite PPI therapy

Exclusion Criteria:

* Extensive esophageal or gastric surgery
* Any chronic illness that would interfere with the study

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Cavallari, PharmD, Principal Investigator — University of Florida; James P Franciosi, MD, Principal Investigator — Nemours Children's Hospital
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Conventional Treatment: For adults randomized to the genotype-supported arm no genotype will be provided to physicians to assist in dosing.
- Pediatric Conventional Treatment: For children randomized to the genotype-supported arm no genotype will be provided to physicians to assist in dosing.
Period: Overall Study
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment
Started | 62 | 63 | 30 | 30
Completed | 56 | 57 | 20 | 23
Not Completed | 6 | 6 | 10 | 7

BASELINE CHARACTERISTICS:
Population: Adult and children ages 5-100 with gastroesophageal reflux disease symptoms expected to take a proton pump inhibitor
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment | Total
Number analyzed (Participants) | 62 | 63 | 30 | 30 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (15.7) | 50.5 (16.3) | 12 (3.7) | 12.5 (3.6) | 39.4 (23.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 17 | 17 | 120
  Male | 19 | 20 | 13 | 13 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 8 | 6 | 25
  Not Hispanic or Latino | 48 | 55 | 22 | 24 | 149
  Unknown or Not Reported | 7 | 4 | 0 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 12 | 7 | 3 | 1 | 23
  White | 46 | 51 | 20 | 27 | 144
  More than one race | 3 | 4 | 6 | 2 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 63 | 30 | 30 | 185

OUTCOME MEASURES:

1. Primary Outcome: Reflux Disease Questionnaire (RDQ)
Description: The RDQ was developed to monitor treatment response over time and evaluates 6 symptoms (12 items) covering 3 domains: heartburn, regurgitation, and upper abdominal pain. Each symptom is evaluated using a 6-point Likert scale to assess frequency and severity over the previous week. Each symptom is rated from 1 (did not have) to 6 (severe), and the RDQ mean score is calculated as the mean response to the 12 items. The RDQ mean score thus ranges from 1 to 6 and has been psycho-metrically validated.
Time Frame: Change from baseline and 12 weeks
Population: Adult patients enrolled that have a CYP2C19 Rapid or Ultra-rapid metabolizer result.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment
Number analyzed (Participants) | 17 | 18 | 0 | 0
score on a scale | -0.387 (1.2) | -0.296 (0.58) |  |
Statistical Analysis 1: Comparison: Adult Genotype Guided Treatment vs Adult Conventional Treatment; We will test the hypothesis that CYP2C19 rapid metabolizers or ultra rapid metabolizers (1 or 2 gain-of-function alleles) in the genotype-supported arm have better gastroesophageal reflux disease and symptom control than CYP2C19 rapid metabolizers or ultra rapid metabolizers in the conventional treatment group because they will have their dose increased based on their genotype; Test type: Superiority — We will test the hypothesis that CYP2C19 rapid metabolizers or ultra rapid metabolizers (1 or 2 gain-of-function alleles) in the genotype-supported arm have better gastroesophageal reflux disease and symptom control than CYP2C19 rapid metabolizers or ultra rapid metabolizers in the conventional treatment group because they will have their dose increased based on their genotype; p = 0.78, t-test, 2 sided — Analysis was done of adult patients enrolled that have a CYP2C19 Rapid or Ultra-rapid metabolizer result

2. Primary Outcome: Pediatric Sinonasal Symptom Survey (SN-5)
Description: The Pediatric Sinonasal Symptom Survey (SN-5) is a validated 5-item scale with each item rated on a scale of worsening symptoms from 1 (none of the time) through 7 (all of the time). Items were averaged to yield a single total score ranging from 1 (better outcomes) to 7 (worse outcomes). The total SN-5 scores were compared between the conventional and genotype-guided dosing groups to determine if one group reported worsening symptoms over the other.
Time Frame: Week 4 (or next available results)
Population: Children aged 5-17 years old with gastric-acid-related conditions and a completed SN-5 questionnaire at week 4 (or next available results)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- Adult Genotype Guided Treatment: For patients randomized to the genotype-supported arm a CYP2C19 genotype will be provided to physicians to assist in dosing.
  CYP2C19 genotyping: All proton pump inhibitors are metabolized in part by the CYP2C19 enzyme, which is encoded by the highly polymorphic CYP2C19 gene. Based on variations within this gene the effectiveness of the drug may be reduced.
- Adult Conventional Treatment: For patients randomized to the genotype-supported arm no genotype will be provided to physicians to assist in dosing.
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment
Number analyzed (Participants) | 0 | 0 | 16 | 18
score on a scale |  |  | 1.8 [1.0 to 2.3] | 2.6 [2.0 to 3.4]
Statistical Analysis 1: Comparison: Pediatric Genotype Guided Treatment vs Pediatric Conventional Treatment; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney) — Adjusted for baseline score, race, baseline proton pump inhibitor use, baseline histamine receptor antagonist use. A sensitivity analysis of participants only on omeprazole revealed similar findings; Adjusted these end points for covariates, including the baseline score, race, and baseline medications using logistic regression

3. Primary Outcome: Safety Questionnaire (SafetyQ)
Description: Occurrence of adverse events over the 12 weeks was captured by the Safety Questionnaire (SafetyQ), which was to be completed on a weekly basis by the parents. The Safety Questionnaire (SafetyQ) asked about the presence of seven different respiratory symptoms since their last visit; upper respiratory infection, sore throat, strep throat, bronchitis, pneumonia, ear infection, and acute sinusitis. If a symptom was selected as being present since the last visit, the date of onset and patient-reported explanation of the symptom was recorded. The number of participants who reported infections were compared between each group.
Time Frame: Over the 12-week period or last date of follow-up
Population: Children aged 5-17 years old with gastric-acid-related conditions with completed SafetyQ assessment over the 12-week period or last date of follow-up
Measure: Number; unit: % of participants reporting infections
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment
Number analyzed (Participants) | 0 | 0 | 26 | 27
% of participants reporting infections |  |  | 20 | 44
Statistical Analysis 1: Comparison: Pediatric Genotype Guided Treatment vs Pediatric Conventional Treatment; Test type: Superiority; p = 0.07, Log Rank — unadjusted; Hazard Ratio (HR) = 2.42, 95% CI 2-sided [0.9 to 6.3]

4. Primary Outcome: Gastroesophageal Reflux Disease (GERD) Assessment of Symptoms in Pediatrics Questionnaire (Gasp-Q)
Description: Gastroesophageal reflux disease (GERD) Assessment of Symptoms in Pediatrics Questionnaire (Gasp-Q) is a validated patient-reported outcome questionnaire that evaluated proton pump inhibitor therapy efficacy. Gasp-Q inquired about the severity and frequency of belly pain, chest pain, difficulty swallowing, choking, burping, nausea, pain after eating, night pain, and vomiting. If the symptom was present, the patient was asked to score the severity of the symptom ranging from 1 (Not at all severe) to 7 (Most severe). A composite score was then calculated based on the scoring of the 9 symptoms and ranged from 9 to 63.
Time Frame: Change in score from baseline to the week 4 ± 1-week
Population: Children aged 5-17 years old with gastric-acid-related conditions and a completed Gasp-Q questionnaire at baseline and week 4 ± 1-week
Measure: Mean (Inter-Quartile Range); unit: median (IQR) composite score
Groups:
- Adult Conventional Treatment: For patients randomized to the genotype-supported arm a no genotype will be provided to physicians to assist in dosing.
- Pediatric Conventional Treatment: For children randomized to the genotype-supported arm a no genotype will be provided to physicians to assist in dosing.
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment
Number analyzed (Participants) | 0 | 0 | 18 | 22
median (IQR) composite score |  |  | -24.0 [-32.0 to -9.0] | -26.0 [-35.0 to 10.0]
Statistical Analysis 1: Comparison: Pediatric Genotype Guided Treatment vs Pediatric Conventional Treatment; If a participant did not complete a follow-up questionnaire during their third to fifth week of proton pump inhibitor therapy, their questionnaire results were excluded from the analyses; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney) — If a participant did not complete a follow-up questionnaire during their third to fifth week of proton pump inhibitor therapy, their questionnaire results were excluded from the analyses

5. Primary Outcome: Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Module
Description: Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Module is a validated patient-reported outcome questionnaire and Likert response scale, to evaluate proton pump inhibitor therapy efficacy. The gastrointestinal problems included in the PedsQL were stomach pain and hurt, stomach upset, food and drink limits, trouble swallowing, heartburn and reflux, gas and bloating, constipation, diarrhea, and worry. Participants were asked to rate the symptoms from 0 (never a problem) to 4 (almost always a problem).
Time Frame: Change in score from baseline to the week 4 ± 1-week
Population: Children aged 5-17 years old with gastric-acid-related conditions with a completed PedsQL questionnaire at baseline and week 4 ± 1-week
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment
Number analyzed (Participants) | 0 | 0 | 19 | 22
score on a scale |  |  | 8.2 [-3.0 to 21.1] | 5.4 [-1.7 to 13.4]
Statistical Analysis 1: Comparison: Pediatric Genotype Guided Treatment vs Pediatric Conventional Treatment; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adult Arms: 24 months after enrollment Pediatric Arms: 12 weeks from baseline
Description: The study was a minimal risk study and all-cause mortality and serious adverse events were not assessed.
Arm/Group | Adult Genotype Guided Treatment | Adult Conventional Treatment | Pediatric Genotype Guided Treatment | Pediatric Conventional Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Pilot study with small sample size and endpoints analyzed in RM/UM subset; no pharmacokinetic analyses done; pragmatic design where any PPI medication could be prescribed; did not account for over-the-counter antacid medications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT02930824/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02930824/ICF_001.pdf